CLINICAL TRIAL: NCT04509791
Title: MELD-ATG: Phase II, Dose Ranging, Efficacy Study of Anti-thymocyte Globulin (ATG) Within 6 Weeks of Diagnosis of Type 1 Diabetes (T1D)
Acronym: Meld-ATG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: S63466; 2019-003265-17 (EudraCT Number)
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum

STUDY DESIGN:
Intervention Model Description: the trial design consists of 7 cohorts, each recruited sequentially, with between 3 and 5 treatment arms ( there will be fewer arms for later cohorts)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- placebo (Placebo Comparator): placebo arm
  Interventions: Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit
- 2.5 mg ATG/kg (Active Comparator): the trial consists of 7 cohorts. The first cohort of 30 participants will be randomised to placebo, 2.5 mg/kg, 1.5 mg/kg, 0.5 mg/kg en 0.1 mg/kg in a 1:1:1:1:1 allocation ratio
  Interventions: Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit
- 1.5 mg ATG/kg (Active Comparator): the next two cohorts of 12 participants will be randomised to placebo, 2.5 mg/Kg, and 2 specified middle ATG total doses in a 1:1:1:1 allocation ratio
  Interventions: Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit
- 0.5 mg ATG/kg (Active Comparator): The next four cohorts of 15 participants will be randomised to placebo, 2.5 mg/kg and a single selected middle ATG total dose in a 1:1:1 allocation ratio
  Interventions: Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit
- 0.1 mg ATG/kg (Active Comparator): the trial consists of 7 cohorts. The first cohort of 30 participants will be randomised to placebo, 2.5 mg/kg, 1.5 mg/kg, 0.5 mg/kg en 0.1 mg/kg in a 1:1:1:1:1 allocation ratio
  Interventions: Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit

INTERVENTIONS:
Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit — MELD - ATG : Minimum effective low dose ant-human thymocyte globulin (rabbit)
  Other Names: ATG

SUMMARY:
This study has been set up within the framework of the INNODIA network. INNODIA is a global partnership between 31 academic institutions, 6 industrial partners, a small sized enterprise and 2 patient organizations, bringing their knowledge and experience together with one common goal: "To fight type 1 diabetes". (www.innodia.eu) The overall aim of INNODIA is to advance in a decisive way how to predict, stage, evaluate and prevent the onset and progression of type 1 diabetes (T1D).

For this, INNODIA has established a comprehensive and interdisciplinary network of clinical and basic scientists, who are leading experts in the field of T1D research in Europe and UK (United Kingdom), with complementary expertise from the areas of immunology, Beta-cell biology, biomarker research and T1D therapy, joining forces in a coordinated fashion with industry partners and two foundations, as well as with all major stakeholders in the process, including regulatory bodies and patients with T1D and their families.

The MELD-ATG trial is a phase II, Multi-centre, randomised, double-blind, placebo-controlled, Multi-arm parallel cohort trial.

* to investigate the effect of 2.5 mg/kg og ATG on the preservation of stimulated C-peptide at 12 months compared to placebo
* to identify the minimally effective dose of ATG that shows an effect on C-peptide when compared to placebo at 12 months

DETAILED DESCRIPTION:
A phase II, Multi-centre, randomised, double-blind, placebo-controlled, Multi-arm parallel cohort trial.

Randomisation wil be stratified by age. The trial consist of seven cohorts. The first cohort of 30 participants will be randomised to placebo, 2.5 mg/kg, 1.5 mg/kg, 0.5 mg/kg and 0.1 mg/kg.

ATG total dose in a 1:1:1:1 allocation ratio. There will be an initial age step down selection of this cohort with recruitment starting with dose aged 12-25 years and, providing no new safety concerns are raised in the first 10 participants to receive active dose, progressing to all ages (5-25 years) The next two cohorts of 12 participants will be randomised to placebo, 2.5 mg/kg, and 2 specified middle ATG total doses in a 1:1:1:1 allocation ratio.

The next four cohorts of 15 participants will be randomised to placebo, 2.5 mg/kg, and a single selected middle ATG total doses in a 1:1:1 allocation ratio.

This design allows sequential adjustment of the middle doses to be explored following review of all safety and early efficacy data by the Independent Data Monitoring Committee ( IDMC) and Dose Determine Committee (DDC) to seek the minimum effective dose

ELIGIBILITY:
Inclusion Criteria:

* has given written informed consent to participate; or have a parent or legal guardian provide written informed consent. Individual under the age of consent will be asked to assent to trial participation
* be aged > 5 years to < 25 years at written informed consent/assent
* have been diagnosed with T1d within 3-9 weeks of planned treatment day 1
* have random C-peptide levels > 200 pmol/L measured at screening, as tested centrally
* have 1 or more diabetes-related autoantibody (GADA, IA-2A or ZnT8A) present at screening, as tested centrally
* will be > 6 weeks form last live immunisation at planned treatment day 1 and be willing to forgo live vaccines during the trial until 6 months post treatment
* be willing to comply with intensive diabetes management

Exclusion Criteria:

* Type 2 diabetes
* Evidence of prior or current tuberculosis (TB) infection
* Clinically significant abnormal full blood count (FBC), renal function or liver function at screening
* Requiring use of other immunosuppressive or immunomodulation agents, including chronic use of systemic steroids
* any active chronic infections at screening, or any active acute or chronic infections at baseline or on treatment day, which would contraindicate any additional immunosuppression
* seropositive for human immunodeficiency virus (HIV),hepatitis B of hepatitis C infection at screening
* positive for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) based on local testing regimen
* unwilling to use appropriate contraception if sexually active during the trial, from date of written informed consent until completion of the 12-month follow-up visit
* any history of malignancies, other than skin
* current or ongoing use of non-insulin pharmaceuticals that effect glycaemic control
* active participation in another T1D treatment interventional trial in the previous 30 days prior to screening ( excluding treatment with insulin)
* any prior treatment with ATG, Abatacept or Anti-CD3 monoclonal antibody (Anti-CD3)
* known allergy to ATG or to similar products
* any condition, complicating medical issues, or abnormal clinical laboratory results that the investigator judges may adversely affect trial conduct, cause increased risk to the participant, or compromise the trial results

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
the area under the stimulated C-peptide response curve | over the first 2 hours of a mixed meal tolerance test (MMTT) at 12 months post treatment

SECONDARY OUTCOMES:
the area under the stimulated C-peptide response curve | over the first 2 hours of a MMTT at baseline, 3, 6 and 12 months
dry blood spot (DBS) C-peptide measurements | at all observation times
Cluster of differentiation 4 (CD4) positive T cells and Cluster of differentiation 8 (CD8) positive T cells | over 12 months
HbA1c | over 12 months
insulin requirements | over 12 months
  The need for insulin (units) on a daily basis
T1D-associated autoantibodies (glutamic acid decarboxylase antibodies (GADA), insulin auto-antibodies (IAA), IA-2 antibodies (IA-2A) and Zinc transporter 8 antibodies (ZnT8A)) | over 12 months
  The presence of T1D-associated autoantibodies
continuous glucose monitoring (CGM) measurements ( time in range, time above time below) | over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: chantal Mathieu, MD,pHD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (14):
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair ziekenhuis Brussel, Brussels
  - Universite Libre de Bruxelles, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Herlev University Hospital, Herlev, Denmark
- Helsinki University Hospital Children and Adolescents, Helsinki, Finland
- Hannoversche Kinderheilanstalt Auf der Bult, Hannover, Germany
- IRCCS Ospedale San Raffaele, Milan, Italy
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- United Kingdom (3):
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxon
  - Cambridge University Hospitals NHS Trust, Cambridge
  - The Royal London Hospital - Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilhelm-Benartzi CS, Miller SE, Bruggraber S, Picton D, Wilson M, Gatley K, Chhabra A, Marcovecchio ML, Hendriks AEJ, Morobe H, Chmura PJ, Bond S, Aschemeier-Fuchs B, Knip M, Tree T, Overbergh L, Pall J, Arnaud O, Haller MJ, Nitsche A, Schulte AM, Mathieu C, Mander A, Dunger D. Study protocol: Minimum effective low dose: anti-human thymocyte globulin (MELD-ATG): phase II, dose ranging, efficacy study of antithymocyte globulin (ATG) within 6 weeks of diagnosis of type 1 diabetes. BMJ Open. 2021 Dec 7;11(12):e053669. doi: 10.1136/bmjopen-2021-053669. PMID 34876434
- [Derived] Mathieu C, Wych J, Hendriks AEJ, Van Ryckeghem L, Tree T, Chmura P, Moller C, Casteels K, Danne T, Reschke F, Smigoc Schweiger D, Battelino T, Johannesen J, Rami-Merhar B, Pieber T, De Block C, Evans M, Hilbrands R, Bosi E, Willemsen RH, Basu S, Pulkkinen MA, Knip M, Cnop M, Nitsche A, Schulte AM, Niemoller E, Peakman M, Wilhelm-Benartzi C, Gillespie D, Overbergh L, Mander AP, Marcovecchio ML; INNODIA. Minimum effective low dose of antithymocyte globulin in people aged 5-25 years with recent-onset stage 3 type 1 diabetes (MELD-ATG): a phase 2, multicentre, double-blind, randomised, placebo-controlled, adaptive dose-ranging trial. Lancet. 2025 Sep 27;406(10510):1375-1388. doi: 10.1016/S0140-6736(25)01674-5. Epub 2025 Sep 18. PMID 40976248